CLINICAL TRIAL: NCT06766734
Title: The Effect of Ultrasound-Guided Tendon Dry Needling on Pain and Function Added to Therapeutic Ultrasound Therapy in Rotator Cuff Tendinopathy
Brief Title: The Effect of Ultrasound-Guided Tendon Dry Needling on Pain and Function in Rotator Cuff Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Berat Bulut, Assistant Doctor, Istanbul Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IstanbulTRH-FTR-BB-01
Record Dates: First submitted 2025-01-04; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: Supraspinatus Tendinopathy
Keywords: Exercise, Supraspinatus tendinopathy, tendinosis, partial tear, dry needling, therapeutic ultrasound, ultrasonography
MeSH Terms: conditions — Motor Activity; Tendinopathy

STUDY DESIGN:
Intervention Model Description: Participants were randomized into 2 groups as a tendon dry needling group or sham tendon dry needling group
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tendon Dry Needling Group (Active Comparator): First tendon dry needling was performed under sterile conditions with real-time imaging guidance using an Esaote MylabFive ultrasound device and a 5-12 MHz linear probe. Then patients were included in an exercise program combined with ultrasound (US) therapy for a total of 15 sessions, 5 times a week for 3 weeks. The second tendon dry needling procedure was performed using the same technique one month after the first tendon dry needling.
  Interventions: Procedure: Tendon Dry Needling
- Sham Tendon Dry Needling Group (Sham Comparator): First sham tendon dry needling was performed under sterile conditions with real-time imaging guidance using an Esaote MylabFive ultrasound device and a 5-12 MHz linear probe. Then patients were included in an exercise program combined with ultrasound (US) therapy for a total of 15 sessions, 5 times a week for 3 weeks. The second sham tendon dry needling procedure was performed using the same technique one month after the first sham tendon dry needling.
  Interventions: Procedure: Sham Tendon Dry Needling

INTERVENTIONS:
Procedure: Tendon Dry Needling — Tendon dry needling procedure is that repetitively passing the needle though the area of supraspinatus tendon. Tendon dry needling was performed under sterile conditions with real-time imaging guidance using an ultrasound probe. The supraspinatus tendon was scanned from anterior to posterior, and tendon dry needling was applied to the identified lesion (tendinozis or partial tear) area. This treatment method was applied twice, with a one-month interval between sessions.
  Arms: Tendon Dry Needling Group
Procedure: Sham Tendon Dry Needling — In this treatment subcutaneous sham tendon dry needling was performed by randomly holding the ultrasound probe in the area corresponding to the same anatomical localization. Sham tendon dry needling performed to subcutaneus tissue not tendon.
  Arms: Sham Tendon Dry Needling Group

SUMMARY:
In this study, we aimed to observe the effect of adding dry needling to therapeutic ultrasound treatment on pain and function in patients with supraspinatus tendinopathy.

DETAILED DESCRIPTION:
One of the common causes of shoulder pain is rotator cuff tendinopathy (RCT). The most affected tendon in RCT is the supraspinatus tendon.

In supraspinatus tendinopathy (SST) various treatment methods are attempted. Conservative treatments are the first-line approach for SST. These include non-steroidal anti-inflammatory drugs (NSAIDs), hot and cold applications, exercise, manual therapy, therapeutic ultrasound (US) therapy, and subacromial steroid injections. Additionally, treatments such as subacromial platelet-rich plasma (PRP) and prolotherapy have been developed. Surgically, rotator cuff repair or subacromial decompression can be performed. Conservative methods can be effective in reducing pain and improving function. While half of shoulder pain cases resolve within 2-3 months, pain persists for more than 12 months in the other half. When we look at the literature, unfortunately there is no gold standard treatment method for SST. Although tendon dry needling is a new treatment method in the treatment of tendinopathy, there are a few articles in the literature about tendon dry needling.

In this study the demographic data (age, gender, occupation (excessive shoulder use (yes/no)), painful shoulder (right, left), dominant hand (right, left), height, weight, body mass index, duration of pain) of the patients who will participate in the study were recorded. Patients were randomized into 2 groups using a closed-envelope method. The first group received DN twice at 4-week intervals under ultrasound guidance (USG) to the supraspinatus tendon, while the second group received placebo DN to a similar anatomical area by randomly positioning the probe. Both groups underwent a total of 15 sessions of US therapy, 5 times a week for 3 weeks, combined with an exercise program. Tendon DN was performed under sterile conditions using an Esaote MylabFive device with a 5-12 MHz superficial probe for real-time imaging in our clinic. To reduce shoulder pain associated with the procedure, 1 ml of 1% prilocaine was injected before the application. A 0.25x40 mm needle was used for DN. In patients who reported pain reduction, the supraspinatus tendon was scanned from front to back, and DN was applied to the detected lesion area. Patients were allowed to continue daily activities, excluding overhead movements, for two weeks. Range of motion (ROM) and Codman shoulder exercises started the day after the injection. Both groups were given progressive resistance supraspinatus strengthening exercises within the pain threshold along with ROM and Codman exercises during the US therapy period. Patient assessments were conducted before treatment, at 1 month (after 15 sessions of therapeutic US treatment and before the 2nd DN), and at 3 months. Patient evaluation parameters included the Visual Analog Scale (VAS) for pain, the Simple Shoulder Test (SST) for function, and SPADI (Shoulder Pain and Disability Index). The evaluator was kept blinded to the treatments provided.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least 6 months of shoulder pain who presented to the outpatient clinic of the Physical Medicine and Rehabilitation Department at SBU Istanbul Training and Research Hospital who agreed to participate in the study.
* Positive examination tests (painful arc, Neer's, Hawkins-Kennedy, Yergason, Speed)
* Positive findings on MRI (tendinosis/partial rupture),

Exclusion Criteria:

* Diagnosis of rheumatologic diseases
* History of intra-articular/subacromial shoulder injection in the last 3 months
* Individuals with a history of shoulder trauma
* Individuals with a history of coronary artery disease
* Cervical origin pain
* Patients with a history of shoulder surgery
* Patients with positive tests for instability
* Patients with a history of humeral fracture
* Diabetes mellitus (DM)
* Patients with adhesive capsulitis
* Individuals allergic to local anesthetic medications
* Full-thickness rotator cuff tear

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-11-10 (Actual); Primary Completion 2024-08-10 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Before treatment, first month, third month
  A tool used to help a person rate the intensity of certain sensations and feelings, such as pain. The visual analog scale for pain is a straight line with one end meaning no pain and the other end meaning the worst pain imaginable. A patient marks a point on the line that matches the amount of pain he or she feels. It may be used to help choose the right dose of pain medicine. Also called VAS.

SECONDARY OUTCOMES:
Shoulder Pain and Disability Index | Before treatment, first month, third month
  The Shoulder Pain and Disability Index (SPADI) was developed to measure current shoulder pain and disability in an outpatient setting. The SPADI contains 13 items that assess two domains; a 5-item subscale that measures pain and an 8-item subscale that measures disability.
Simple Shoulder Test | Before treatment, first month, third month
  Simple Shoulder Test The SST is a self-reported shoulder-specific questionnaire that measures functional limitations of the affected shoulder in patients with shoulder dysfunction.18 The SST consists of 12 questions with dichotomous (yes/ no) response options.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Training and Research Hospital, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR